CLINICAL TRIAL: NCT03295084
Title: Irinotecan Gastro-resistant Tablet. An Open Label Phase I, Dose Escalating Study Evaluating Safety, Tolerability and Pharmacokinetics of Oral Administration of Irinotecan in Adult Patients With Solid Tumors
Brief Title: Safety, Tolerability and Pharmacokinetics of Oral Tablet of Irinotecan in Adult Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dorte Nielsen (Other)
Responsible Party: Sponsor-Investigator, Dorte Nielsen, Professor, MD, DMSci, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AA1446
Record Dates: First submitted 2017-09-11; First posted 2017-09-27 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; Capecitabine

STUDY DESIGN:
Intervention Model Description: Open labelled study with enrollment in the order of confirmation of eligibility. Escalating doses of study drug in sequential patient cohorts for identification of DLT and MTD (Phase 1)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Irinotecan (Experimental): Dose escalation study in cohorts of minimum 3 patients of an Irinotecan tablet taken once daily for 14 days within 3 week treatment cycle
  Interventions: Drug: Irinotecan
- Irinotecan with Capecitabine (Experimental): Dose escalation study in cohorts of minimum 3 patients of an Irinotecan tablet taken once daily in combination with Capecitabine tablet taken twice daily for 14 days within 3 week treatment cycle
  Interventions: Drug: Irinotecan; Drug: Capecitabine

INTERVENTIONS:
Drug: Irinotecan — Dose Escalation
Drug: Capecitabine — Dose Escalation
  Arms: Irinotecan with Capecitabine

SUMMARY:
This study evaluates the safety, tolerability and pharmacokinetics of oral administration of irinotecan in adult patients. Oral irinotecan will be administered as monotherapy in a dose escalation trial to establish the Maximal Tolerated Dose. Totally 25 patients will be treated with irinotecan tablets as mono-therapy. As an extension trial 12 patients will be treated with oral irinotecan in combination with oral capecitabine

DETAILED DESCRIPTION:
The study is a phase I, open-label, dose escalation single center study in patients with solid tumors. The study will investigate safety, tolerability and Maximal Tolerated Dose as primary end-points of an irinotecan tablet given as single agent or in combination with oral capecitabine. Secondary end-points are pharmacokinetics and preliminary anti-tumor response.

Cohorts of 3 patients will be treated on selected dose level with oral irinotecan in order to identify Dose Limiting Toxicity (DLT) and Maximal Tolerated Dose (MTD). Totally 12 subjects will be treated at the MTD level. Patients will receive irinotecan tablets once daily in the morning for 14 consecutive days within 3 week treatment cycles. As an extension trial totally 12 subjects will be treated with oral irinotecan in combination with oral capecitabine. Patients treated in combination therapy will receive irinotecan tablets once daily in the morning for 14 consecutive days in combination with capecitabine dosed twice daily for 14 consecutive days within 3 week treatment cycles.

ELIGIBILITY:
Inclusion Criteria:

* Signed written Informed Consent
* 18 years of age or older
* Capable of understanding the protocol requirements and risk associated with the study
* Patients must have histological confirmed malignancy (solid tumor) that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
* Patients with either measurable disease according to RECIST 1.1 or non-measurable disease
* Performance status 0-1 (ECOG)
* Life expectancy ≥ 3 months
* Coagulation INR < 1.3 and APTT within normal limits
* WBC ≥ 3000/mm3
* Absolute neutrophil count ≥ 1500/mm3
* Hemoglobin ≥ 6.0 mmol/L
* Platelet count ≥ 100.000/mm3
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN AST and ALT ≤ 2.5 times ULN. For patients with liver metastasis adequate hepatic function is defined by aspartate aminotransferase (AST) ≤ 5 x ULN and alanine aminotransferase ALT ≤ 5 x ULN
* No severe or uncontrolled renal condition (creatinine ≤ than 1.5 ULN)
* No significant cardiovascular disease (New York Heart Association Class III and IV)
* No other severe cardiac condition not defined above
* No significant cardiovascular disease (incl. myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) ≤ 1 year prior for patients to be enrolled and treated in combination with oral capecitabine
* No severe or uncontrolled pulmonary condition
* No known prior hypersensitivity reaction to irinotecan
* No known prior hypersensitivity to capecitabine or 5-fluorouracil for patients to be enrolled and treated in combination with oral capecitabine
* No chronic enteropathy (e.g. active inflammatory bowel disease, extensive intestinal resection or chronic diarrhea)
* No bowel obstruction or sub-obstruction
* No prior history of intestinal malabsorption
* Patients have to be able to swallow normally and have to be willing to comply with the intake of tablets
* No psychiatric condition that would preclude study participation
* No co-existing active infection requiring antibiotics or any co-existing medical conditions likely to interfere with study procedures
* No other condition that will preclude study participation
* A negative pregnancy test for women of childbearing potential. For men and women of child-producing potential, the use of effective contraceptives methods during the study and at least 3 months after discontinuations of the study drug is required.
* Not pregnant or nursing
* Peripheral neuropathy NCI CTCAE grade less than 2 for patients to be enrolled and treated in combination with oral capecitabine
* The patient is willing and able to comply with hospitalization for treatment and scheduled follow-up visits and examinations

Exclusion Criteria:

* Simultaneous participation in any other study involving investigational drugs or having participated in a study within 4 weeks prior to start of study treatment
* Symptomatic brain metastases
* Intake of any prohibited concomitant medication
* Known Dihydropyrimidine dehydrogenase (DPD) deficiency for patients to be enrolled and treated in combination with oral capecitabine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-07-15 (Actual); Primary Completion 2018-07-03 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Maximal Tolerated Dose (MTD) and Dose Limiting Toxicity (DLT) of oral Irinotecan based on incidence of Treatment-Emergent Adverse Events | 2 treatment cycles of 3 weeks
  Number of patients with Treatment Related Adverse Events as assessed according to the NCI Common Terminology Criteria for Adverse events CTCAE version 4.0

SECONDARY OUTCOMES:
Maximum Tolerated Dose (MTD) and the Dose Limiting Toxicity (DLT) of oral Irinotecan in combination with oral Capecitabine based on incidence of Treatment-Emergent Adverse Events | 2 treatment cycles of 3 weeks
  Number of patients with Treatment Related Adverse Events as assessed according to the NCI Common Terminology Criteria for Adverse events CTCAE version 4.0
Area under the Concentration-Time-Curve (AUC) for Irinotecan and its metabolites SN-38 and SN-38 glucoronide | Day 1 and Day 14 of first 3 weeks treatment cycle
  PK samples will be collected at predetermined time intervals and pharmacokinetic parameter calculated and reported based on the plasma concentration profile
Maximum Serum Concentration (Cmax) for irinotecan and its metabolites SN-38 and SN-38 glucoronide | Day 1 and Day 14 of first 3 weeks treatment cycle
  PK samples will be collected at predetermined time intervals and pharmacokinetic parameter calculated and reported based on the plasma concentration profile
Time to Maximum Serum Concentration (Tmax) for irinotecan and its metabolites SN-38 and SN-38 glucoronide | Day 1 and Day 14 of first 3 weeks treatment cycle
  PK samples will be collected at predetermined time intervals and pharmacokinetic parameter calculated and reported based on the plasma concentration profile
Half-life (t½) for irinotecan and its metabolites SN-38 and SN-38 glucoronide | Day 1 and Day 14 of first 3 weeks treatment cycle
  PK samples will be collected at predetermined time intervals and pharmacokinetic parameter calculated and reported based on the plasma concentration profile
Serum concentration 24 hours after dosing and prior to administration of the next dose (C24) for Irinotecan and its metabolites SN-38 and SN-38 glucoronide | Day 1 and Day 14 of first 3 weeks treatment cycle
  PK samples will be collected at predetermined time intervals and pharmacokinetic parameter calculated and reported based on the plasma concentration profile
Objective tumor response to treatment based on RECIST 1.1 criteria | 2 treatment cycles of 3 weeks
  CT scans with tumor response as assessed using RECIST 1.1. criteria

CONTACTS AND LOCATIONS:
Overall Officials: Benny Vittrup, Principal Investigator — Herlev Hospital, Department of Oncology, Denmark
Locations (1):
- Herlev Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: Undecided